CLINICAL TRIAL: NCT00654589
Title: A One-year, Open-label, Single Arm, Multi-center Trial Evaluating the Efficacy and Safety of Oral ICL670 (20 mg/kg/d) in Patients Three to Six Months After Allogeneic Hematopoietic Cell Transplantation in Whom Iron Overload is Present
Brief Title: Efficacy and Safety of Oral Deferasirox (20 mg/kg/d) in Pts 3 to 6 Months After Allogeneic Hematopoietic Cell Transplantation Who Present With Iron Overload
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670ADE02
Record Dates: First submitted 2008-04-02; First posted 2008-04-08 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Iron Overload
Keywords: Hematopoietic stem cell transplantation; HCT; iron overload; chelators; ICL670; deferasirox; serum ferritin; LIC; transfusional hemosiderosis; blood transfusions; adults; iron chelation; 3-6 months; allogeneic hematopoietic stem cell transplantation
MeSH Terms: conditions — Iron Overload | interventions — Deferasirox

ARMS (1):
- deferasirox (Experimental)
  Interventions: Drug: Deferasirox

INTERVENTIONS:
Drug: Deferasirox
  Other Names: ICL670

SUMMARY:
The purpose of this study is to investigate the effects of iron chelation using deferasirox in patients who show signs of iron overload after an allogeneic stem cell transplantation The iron overload must be due to blood transfusions.

ELIGIBILITY:
Inclusion criteria:

1. Transfusional iron overload three to six months after HCT with no evidence of active inflammation
2. History of at least 20 units of red blood cell transfusions or 100mL/kg of prepacked red blood cells (PRBCs).
3. Patients of either gender and age ≥ 18 years.
4. Female patients who have reached menarche and who are sexually active must use double-barrier contraception, oral contraceptive plus barrier contraception , or must have undergone clinically documented total hysterectomy and/or ovariectomy, or tubal ligation or be postmenopausal defined by amenorrhea for at least 12 months.

Exclusion criteria:

1. Non-transfusion related iron overload
2. Active malignancy
3. Known active viral hepatitis or known HIV positiveness
4. Mean levels of alanine aminotransferase (ALT) > 5x ULN
5. Treatment with any iron chelator after transplantation
6. Uncontrolled systemic hypertension
7. Serum creatinine > 1.5 ULN and/or serum creatinine clearance < 60 ml/min
8. History of nephrotic syndrome.
9. Previous history of clinically relevant ocular or auditory toxicity related to iron chelation.
10. Systemic diseases (cardiovascular, renal, hepatic, etc.) which would prevent the patient from undergoing study treatment
11. Pregnant or breast feeding patients.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2008-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
To assess iron chelation by comparing serum ferritin values at baseline vs. 52 weeks of treatment with deferasirox | 52 weeks

SECONDARY OUTCOMES:
To evaluate the relationship between serum ferritin, transferrin (TRF) and transferrin saturation during the whole study. | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (1):
- Novartis Investigative Site, Leipzig, Germany

REFERENCES:
- [Result] Jaekel N, Lieder K, Albrecht S, Leismann O, Hubert K, Bug G, Kroger N, Platzbecker U, Stadler M, de Haas K, Altamura S, Muckenthaler MU, Niederwieser D, Al-Ali HK. Efficacy and safety of deferasirox in non-thalassemic patients with elevated ferritin levels after allogeneic hematopoietic stem cell transplantation. Bone Marrow Transplant. 2016 Jan;51(1):89-95. doi: 10.1038/bmt.2015.204. Epub 2015 Sep 14. PMID 26367238